CLINICAL TRIAL: NCT04398589
Title: The Effect of Dexmedetomidine for Suprascapular Nerve Block With Axillary Nerve Block on Plasma Cortisol and Pain-related Cytokines After Arthroscopic Rotator Cuff Repair: a Randomized Controlled Trial
Brief Title: The Effect of Dexmedetomidine for Suprascapular Nerve Block With Axillary Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Hallym University (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Associate Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-20
Record Dates: First submitted 2020-05-08; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Suprascapular Nerve Block; Axillary Nerve Block; Dexmedetomidine; Arthroscopic Rotator Cuff Repair; Postoperative Pain; Pain Related Cytokine
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSNB and ANB c DEX (Experimental): We used 9.5 ml of 0.75% ropivacaine and 0.5 ml (50 μg) of dexmedetomidine each for SSNB and ANB.
  Interventions: Drug: Dexmedetomidine injection
- SSNB and ANB c saline (Placebo Comparator): We used 9.5 ml of 0.75% ropivacaine and 0.5 ml normal saline each for SSNB and ANB.
  Interventions: Drug: Saline injection

INTERVENTIONS:
Drug: Dexmedetomidine injection — We used 9.5 ml of 0.75% ropivacaine and 0.5 ml (50 μg) of dexmedetomidine each for preemptive suprascapular nerve block and axillary nerve block just before arthroscopic repair of rotator cuff tear.
  Other Names: suprascapular nerve block and axillary nerve block c ropivacaine; arthroscopic rotator cuff repair
  Arms: SSNB and ANB c DEX
Drug: Saline injection — We used 9.5 ml of 0.75% ropivacaine and 0.5 ml normal saline each for preemptive suprascapular nerve block and axillary nerve block just before arthroscopic repair of rotator cuff tear.
  Other Names: suprascapular nerve block and axillary nerve block c ropivacaine; arthroscopic rotator cuff repair
  Arms: SSNB and ANB c saline

SUMMARY:
Suprascapular nerve block (SSNB) is most commonly used for relieving postoperative pain of arthroscopic rotator cuff repair and it can be used in combination with axillary nerve block (ANB). Dexmedetomidine (DEX) is known as a type of alpha agonist which can elongate the duration of regional block. The aim of this study was to compare the results of dexmedetomidine combined with SSNB and ANB with SSNB and ANB alone on postoperative pain, satisfaction, and pain-related cytokines within the first 48 hours after arthroscopic rotator cuff repair.

Forty patients with rotator cuff tears who had undergone arthroscopic rotator cuff repair were enrolled in this single center, double-blinded randomized controlled trial study. Twenty patients were randomly allocated to group 1 and received ultrasound-guided SSNB and ANB using each mixture of 0.5 ml (50 μg) of DEX and 9.5 ml of 0.75% ropivacaine preemptively. The other 20 patients were allocated to group 2 and underwent ultrasound-guided SSNB and ANB alone using a mixture of 0.5 ml of normal saline and 9.5 ml of ropivacaine. The visual analog scale (VAS) for pain and patient satisfaction (SAT) scores were checked within 48 h postoperatively. The plasma interleukin (IL)-6, -8,-1β, cortisol, and serotonin levels were also measured within 48 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* defined rotator cuff tear on preoperative MRI, which indicated repair
* acceptable arthroscopic surgery, including rotator cuff repair
* patients >20 years old
* acceptable routine regional blocks and patient-controlled analgesia (PCA)

Exclusion Criteria:

* did not undergo arthroscopic rotator cuff repair
* stopped PCA before 48 h postoperatively due to side effects
* had a concomitant operation for a Bankart lesion
* had a history of shoulder operation or fracture
* had a concomitant neurological disorder around the shoulder
* underwent conversion to open surgery from the arthroscopy
* had contraindications for the routine regional blocks used in this study
* had an known allergy or hypersensitivity against ropivacaine or dexmedetomidine, including other amino-amide local anesthetics or α2-adrenoceptor agonists.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale of pain | change from baseline VAS pain score at hour 48
  The VAS pain score was based on a scale from 0 to 10, where 0 indicated no pain and 10 indicated severe pain.

SECONDARY OUTCOMES:
patient's satisfaction | change from baseline patient's satisfaction score at hour 48
  patient's satisfaction score was based on a scale from 0 to 10, where 0 indicated no satisfaction and 10 indicated much satisfaction.
Plasma cortisol level | change from baseline plasma cortisol level at hour 48
  A 3-ml blood sample was retrieved from the peripheral vein of the contralateral upper limb or both lower limbs per sampling.
Plasma IL-6 level | change from baseline plasma IL-6 level at hour 48
  A 3-ml blood sample was retrieved from the peripheral vein of the contralateral upper limb or both lower limbs per sampling.
Plasma IL-8 level | change from baseline plasma IL-8 level at hour 48
  A 3-ml blood sample was retrieved from the peripheral vein of the contralateral upper limb or both lower limbs per sampling.
Plasma IL-1β level | change from baseline plasma IL-1β level at hour 48
  A 3-ml blood sample was retrieved from the peripheral vein of the contralateral upper limb or both lower limbs per sampling.
Plasma serotonin level | change from baseline plasma serotonin level at hour 48
  A 3-ml blood sample was retrieved from the peripheral vein of the contralateral upper limb or both lower limbs per sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Study Chair — Chuncheon Sacred Heart Hospital, Hallym University Medical College
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
We will discuss it with our IRB.

REFERENCES:
- [Derived] Lee JJ, Kim DY, Hwang JT, Song DK, Lee HN, Jang JS, Lee SS, Hwang SM, Moon SH, Shim JH. Dexmedetomidine combined with suprascapular nerve block and axillary nerve block has a synergistic effect on relieving postoperative pain after arthroscopic rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4022-4031. doi: 10.1007/s00167-020-06288-8. Epub 2020 Sep 25. PMID 32975624